CLINICAL TRIAL: NCT04997590
Title: Clinical Study of Umbilical Cord Blood Mononuclear Cells (UCB-MNCs) in Promoting Traumatic Fracture Healing
Brief Title: Clinical Study of Umbilical Cord Blood Mononuclear Cells (UCB-MNCs) in the Treatment of Traumatic Fracture Healing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qianfoshan Hospital (Other)
Collaborators: Shandong Qilu Stem Cells Engineering Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Lili Cao, Professor, Qianfoshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YXLL-KY-2020(041)
Record Dates: First submitted 2021-07-26; First posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Bone Nonunion
Keywords: Umbilical cord blood mononuclear cells; Traumatic fracture healing; Bone nonunion
MeSH Terms: interventions — enterotoxin C, staphylococcal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Umbilical cord blood mononuclear cells group (Experimental): Umbilical cord blood mononuclear cells (cell number 1×108/2mL), once every two weeks, 3 times in total.
  Interventions: Biological: Umbilical cord blood mononuclear cells
- Staphylococcal Enterotoxin C group (Active Comparator): Staphylococcal enterotoxin C (2mL), once every two weeks, 3 times in total.
  Interventions: Drug: Staphylococcal Enterotoxin C

INTERVENTIONS:
Biological: Umbilical cord blood mononuclear cells — injection of CB-MNCs (cell count 1×108 cells/time) was performed once every 2 week for a total of 3 times.
  Arms: Umbilical cord blood mononuclear cells group
Drug: Staphylococcal Enterotoxin C — injection of staphylococcal enterotoxin C was performed once every 2 week for a total of 3 times.
  Arms: Staphylococcal Enterotoxin C group

SUMMARY:
The aim of this study is to explore the effectiveness and safety of umbilical cord blood mononuclear cells in promoting traumatic fracture healing.

DETAILED DESCRIPTION:
Umbilical cord blood mononuclear cells are a type of cell group containing hematopoietic stem cells, mesenchymal stem cells, neural stem cells, endothelial cells, immune cells, etc.In this study ,umbilical cord blood mononuclear cells will be used in promoting traumatic fracture healing,and the effectiveness and safety of the treatment plan was evaluated by twelve months of follow-up after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic long bone fracture.
* Noninfectious bone nonunion, delayed bone union.
* 3 months after the operation of the fracture, the examination showed no callus growth, no signs of progressive repair at the fracture site, fracture piece space < 5mm.
* No shortening, angulation and displacement.
* There was no obvious callus growth 8 months after local bone grafting.

Exclusion Criteria:

* There are infection foci at and near the fracture end after fracture.
* 3 months after the fracture, tests showed partial callus growth.
* Combining shortening, angulation and displacement phenomena.
* Partial callus grew 8 months after local bone grafting.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-12-10 (Actual); Primary Completion 2021-12-10 (Estimated); Study Completion 2022-12-10 (Estimated)

PRIMARY OUTCOMES:
Bone formation | 1 month to 1 year after treatment
  If there is no bone formation, 0 points. Bone formation accounts for 25% of the fracture area, 1 point. Bone formation accounts for 50% of the fracture area, 2 points. Bone formation accounts for 75% of the fracture area, 3 points. Bone filled the gap between fracture ends, 4 points.
Bone defect connection | 1 month to 1 year after treatment
  0 points for complete fracture lines, 2 points for partial fracture lines, 4 points for lack of fracture lines.
Bone reconstruction | 1 month to 1 year after treatment
  0 points for no manifestations of reconstruction,2 points for intramedullary cavity can be reconstructed , and 4 points for the cortical bone can be completely reconstructed. A total score of 11 points or more achieves a good healing effect.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Liang, doctor, Principal Investigator — Qianfoshan Hospital
Locations (1):
- China, Shandong Qianfoshan Hospital, Jinan, Shandong, China